CLINICAL TRIAL: NCT05687383
Title: The Effect of Modified Pillow on Safety During Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: N202210042
Record Dates: First submitted 2023-01-04; First posted 2023-01-18 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2022-12

CONDITIONS: Breastfeeding; Pregnancy Related; Newborn; Fit; Safety Issues
Keywords: Breastfeeding; Pillow; Safety issues; Comfort; Newborn; Pregnancy
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safe breastfeeding pillow (Experimental): Safe breastfeeding pillow increase the comfort and safety of postpartum women during breastfeeding, thereby prolonging breastfeeding and ensuring optimal nutrition for the baby
  Interventions: Device: Safe breastfeeding pillow
- Breastfeeding pillow (Placebo Comparator): Providing a comfortable, supportive and safe environment for healthier and breastfeeding for women and babies
  Interventions: Device: Safe breastfeeding pillow

INTERVENTIONS:
Device: Safe breastfeeding pillow — A randomized controlled trial
  Other Names: Breastfeeding pillow

SUMMARY:
This study will investigate the effectiveness of a modified product "safe breastfeeding pillow" in enhancing the comfort and safety of postpartum women during breastfeeding. The results of this study can be used as a reference to promote clinical practice and education on breastfeeding to prolong the duration of breastfeeding and to ensure the safety of newborns.

DETAILED DESCRIPTION:
Breastfeeding has a significant long-term positive impact on the health, nutrition and development of children, as well as the physical and mental health of women. Baby-Friendly Hospital Initiative (BFHI) was launched by the World Health Organization and UNICEF in 1991 to encourage comfortable, supportive, and safe breastfeeding environments (Byrom et al., 2021). During breastfeeding, mothers need to maintain the same position with their hands for long periods of time, which can lead to muscle pain due to improper posture. In addition, postpartum fatigue can also lead to newborn fall accidents (Lipke et al., 2018).

Objective: To investigate the effectiveness of a modified pillow to enhance the comfort and safety of postpartum women during breastfeeding.

METHODS: A randomized controlled trial was conducted. Mothers and infants who gave birth naturally without serious postpartum complications at a university affiliate hospital will recruit in northern Taiwan. A questionnaire containing "Breastfeeding Self-Efficacy Scale (BSES)", "B-R-E-A-S-T-Feed scale", "Breastfeeding safety scale", and "Body Part Discomfort Scale (BPDS)" will be used to assess comfort and safety during breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

1. Normal spontaneous delivered mothers without serious postpartum complications.
2. Normal newborns who can breastfeed.
3. The mother is willing to breastfeed at least 3 times in the cradle position during the hospital stay.
4. Mothers can communicate in Chinese and Taiwanese.
5. Agree to participate in the study and complete the informed consent form.

Exclusion Criteria:

1. Infants who cannot continue breastfeeding due to condition changes after birth.
2. Mothers who cannot continue breastfeeding due to medical reasons after childbirth.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 150 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Breastfeeding Self-Efficacy Scale (BSES) | through study completion, an average of 2-7 days
  A 14-item self-administered instrument derived from the original 33-item BSES that measures breastfeeding confidence

SECONDARY OUTCOMES:
Breastfeeding safety scale | through study completion, an average of 2-7 days
  A total of four questions using "The Likert scale" to evaluate the mother's level of safety during breastfeeding using a 4-point, with 1 point indicating "very worrying" and 4 points representing "very secure."
Body Part Discomfort Scale (BPDS) | through study completion, an average of 2-7 days
  Used to evaluate the comfort level of body parts during breastfeeding of parturients. There are 10 items in total, and the 4-point Likert scale is used for scoring, with 1 point representing "very uncomfortable" and 4 points representing "very comfortable".
B-R-E-A-S-T-Feed scale | through study completion, an average of 2-7 days
  Evaluate the breastfeeding position and latching position of the parturient. The evaluation items include: Body position, responses, emotional bonding, anatomy, suckling, time spent sucking

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan